CLINICAL TRIAL: NCT04702698
Title: Phase I, Open-Label, Randomized, Single-Dose Study With Crossover Design to Investigate the Effect of Food on the PK of Peposertib Tablet Formulation and to Investigate the PK of Peposertib Administered as Oral Suspension of Disintegrated Tablets
Brief Title: Effect of Food on Peposertib PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS100036_0040; 2020-004187-26 (EudraCT Number)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: Peposertib; Pharmacokinetics; Relative Bioavailability
MeSH Terms: interventions — peposertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part 1: Peposertib: Treatment Sequence A-B-C (Experimental): Participants will receive single oral dose of peposertib tablet (Treatment A) on Day 1 under fasted condition in period 1, followed by single oral dose of peposertib tablet (Treatment B) on Day 8 under fed condition in period 2, followed by oral suspension dose of peposertib (Treatment C) on Day 15 under fasted condition in period 3. There will be washout period of 7 days between each treatment period.
  Interventions: Drug: Peposertib
- Part 1: Peposertib Treatment Sequence A-C-B (Experimental): Participants will receive single oral dose of peposertib tablet (Treatment A) on Day 1 under fasted condition in period 1, followed by oral suspension dose of peposertib (Treatment C) on Day 8 under fasted condition in period 2, followed by single oral dose of peposertib tablet (Treatment B) on Day 15 under fed condition in period 3. There will be washout period of 7 days between each treatment period.
  Interventions: Drug: Peposertib
- Part 1: Peposertib Treatment Sequence B-A-C (Experimental): Participants will receive single oral dose of peposertib tablet (Treatment B) on Day 1 under fed condition in period 1, followed by single oral dose of peposertib tablet (Treatment A) on Day 8 under fasted condition in period 2, followed by oral suspension dose of peposertib (Treatment C) on Day 15 under fasted condition in period 3. There will be washout period of 7 days between each treatment period.
  Interventions: Drug: Peposertib
- Part 1: Peposertib Treatment Sequence B-C-A (Experimental): Participants will receive single oral dose of peposertib tablet (Treatment B) on Day 1 under fed condition in period 1, followed by oral suspension dose of peposertib (Treatment C) on Day 8 under fasted condition in period 2, followed by single oral dose of peposertib tablet (Treatment A) on Day 15 under fasted condition in period 3. There will be washout period of 7 days between each treatment period.
  Interventions: Drug: Peposertib
- Part 1: Peposertib: Treatment Sequence C-A-B (Experimental): Participants will receive oral suspension dose of peposertib (Treatment C) on Day 1 under fasted condition in period 1, followed by single oral dose of peposertib tablet (Treatment A) on Day 8 under fasted condition in period 2, followed by single oral dose of peposertib tablet (Treatment B) on Day 15 under fed condition in period 3. There will be washout period of 7 days between each treatment period.
  Interventions: Drug: Peposertib
- Part 1: Peposertib Treatment Sequence C-B-A (Experimental): Participants will receive oral suspension dose of peposertib (Treatment C) on Day 1 under fasted condition in period 1, followed by single oral dose of peposertib tablet (Treatment B) on Day 8 under fed condition in period 2, followed by single oral dose of peposertib tablet (Treatment A) on Day 15 under fasted condition in period 3. There will be washout period of 7 days between each treatment period.
  Interventions: Drug: Peposertib
- Part 2: Peposertib Treatment Sequence A-B (Experimental): Participants will receive single oral dose of peposertib tablet (Treatment A) on Day 1 under fasted condition in period 1, followed by single oral dose of peposertib tablet (Treatment B) on Day 8 under fed condition in period 2. There will be washout period of 7 days between each treatment period.
  Interventions: Drug: Peposertib
- Part 2: Peposertib: Treatment Sequence B-A (Experimental): Participants will receive single oral dose of peposertib tablet (Treatment B) on Day 1 under fed condition in period 1, followed by single oral dose of peposertib tablet (Treatment A) on Day 8 under fasted condition in period 2. There will be washout period of 7 days between each treatment period.
  Interventions: Drug: Peposertib

INTERVENTIONS:
Drug: Peposertib — Participants will receive single oral dose of Peposertib tablet under fasting (Treatment A) or fed (Treatment B) conditions.
  Other Names: MSC2490484A; M3814
Drug: Peposertib — Participants will receive oral suspension dose of peposertib tablets under fasted condition (Treatment C) in either period 1, 2 or 3 of part 1.
  Other Names: MSC2490484A; M3814
  Arms: Part 1: Peposertib Treatment Sequence A-C-B; Part 1: Peposertib Treatment Sequence B-A-C; Part 1: Peposertib Treatment Sequence B-C-A; Part 1: Peposertib Treatment Sequence C-B-A; Part 1: Peposertib: Treatment Sequence A-B-C; Part 1: Peposertib: Treatment Sequence C-A-B

SUMMARY:
The study will investigate the effect of food on the Pharmacokinetic (PK) of a single dose of peposertib administered as film-coated tablet under fed and fasted conditions. Furthermore, the PK profile of peposertib administered as an oral suspension of disintegrated tablets and as film-coated tablets will be compared under fasted conditions to evaluate the relative bioavailability in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring
* Participants are nonsmoker for at least 6 months prior to Screening
* Participants have a body weight greater than 50 kilogram (kg) and a body mass index within the range 18.5 to 30.0 kilogram per meter square (inclusive) at Screening
* Male participants are refrain from donating sperm plus either abstain from any activity that allows for exposure to ejaculate
* Female participants are not pregnant or breastfeeding
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History of clinically relevant renal, cardiovascular, pulmonary disease, or endocrinology disorder at Screening
* History of clinically relevant gastrointestinal disease, in particular pancreatic disease, cholecystitis, liver diseases or hepatic dysfunction at Screening
* History of psychiatric or relevant neurological disorders (example, depression, epilepsy) at Screening
* History of relevant skin and mucosal diseases (rash, mucositis) at Screening
* Presence or history of any serious allergy (requiring hospitalization or prolonged systemic treatment) at Screening
* Any planned radiologic assessments during the study conduct phase
* Participants who are not able or willing to eat the entire study meals.
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Sampling (AUC0-tlast) of Peposertib | Pre-dose up to 36 hours post-dose
Part 1 and Part 2: Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUC-inf) of Peposertib | Pre-dose up to 36 hours post-dose
Part 1 and Part 2: Maximum Observed Plasma Concentration (Cmax) of Peposertib | Pre-dose up to 36 hours post-dose

SECONDARY OUTCOMES:
Part 1 and Part 2: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs | Part 1: up to 21 days; Part 2: up to 14 days
Part 1 and Part 2: Number of Participants With Treatment -Emergent Adverse Events (TEAEs) Based on Severity According to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | Part 1: up to 21 days; Part 2: up to 14 days
Part 1 and Part 2: Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters, Vital Signs and 12-Lead Electrocardiogram (ECG) Findings | Part 1: up to 21 days; Part 2: up to 14 days
  Number of participants with clinically significant change from baseline in laboratory parameters, vital signs and 12-Lead electrocardiogram (ECG) findings will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (2):
- Germany (2):
  - Nuvisan GmbH, Gauting
  - Nuvisan GmbH, Neu-Ulm

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany, will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.merckgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- [Derived] Becker A, Krebs-Brown A, Vetter C, Reuter T, Rodriguez-Gutierrez A, You X, Lissy M. Phase I crossover study of DNA-protein kinase inhibitor peposertib in healthy volunteers: Effect of food and pharmacokinetics of an oral suspension. Clin Transl Sci. 2023 Dec;16(12):2628-2639. doi: 10.1111/cts.13657. Epub 2023 Oct 31. PMID 37905356
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS100036_0040
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html